CLINICAL TRIAL: NCT06404580
Title: The Benefits of R Anastomotic Technique for Billroth-II Reconstruction With Braun Anastomosis During Totally Laparoscopic Distal Gastrectomy: a Propensity Score Matching Analysis
Status: Completed | Type: Observational
Sponsor: Daorong Wang (Other)
Responsible Party: Sponsor-Investigator, Daorong Wang, DR, Northern Jiangsu People's Hospital
Organization: Northern Jiangsu People's Hospital (Other)
Other Study IDs: R vs B-II-B
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: the Incidences of Clavien-Dindo Grade II or Higher; Anastomotic Time

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- R anastomosis
  Interventions: Procedure: R anastomosis
- B-II-B anastomosis
  Interventions: Procedure: R anastomosis

INTERVENTIONS:
Procedure: R anastomosis — R anastomosis

SUMMARY:
Between March 2019 and September 2022 in our centre, R anastomosis was performed on 123 patients undergoing TLDG for distal gastric cancer. A retrospective review of a prospectively collected database identified patients who underwent TLDG between January 2010 and September 2022. Patients who underwent R anastomosis were matched in a 1:1 ratio with patients who underwent conventional anastomosis using a propensity score based on age, sex, preoperative BMI, American Society of Anesthesiologists (ASA) score, and the history of abdominal surgery. Surgical and postoperative outcomes and clinicopathological data were analyzed for both groups.

ELIGIBILITY:
Inclusion Criteria:

1. elective surgery for endoscopic and pathological diagnosis of malignant tumour of the gastric antrum or body with no distant metastases confirmed by multilayer spiral computed tomography;
2. patients who underwent B-II-B anastomosis during TLDG; and (3) patients who could be followed up postoperatively.

Exclusion Criteria:

(1) patients who had received preoperative neoadjuvant radiotherapy or chemotherapy; (2) patients undergoing emergency surgery; (3) the presence of other malignant tumours concurrently; and (4) patients who were lost to follow-up.

Ages: 35 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: between March 2019 and September 2022 at Northern Jiangsu people's hospital were prospectively collected, and data from patients who underwent conventional anastomosis (control group) were retrospectively collected from the same prospectively maintained database of patients who underwent TLDG between January 2010 and February 2019 at Northern Jiangsu people's hospital.
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
the incidences of Clavien-Dindo grade II or higher | 2010-2022
  the incidences of Clavien-Dindo grade II or higher
anastomotic time | 2010-2022
  anastomotic time

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Jiangsu People's Hospital, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No